CLINICAL TRIAL: NCT04593667
Title: Utilizing a Novel Agent in a Randomized Study of Accelerated Radial Arterial Hemostasis Under Reduced Compression Following Percutaneous Transradial Coronary Angiography/Intervention
Brief Title: Randomized Study of Accelerated Radial Arterial Hemostasis
Acronym: GOLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medcura Inc. (Industry)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WIRB Protocol 20202766; 1291856 (Other: WIRB)
Record Dates: First submitted 2020-10-07; First posted 2020-10-20 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2020-10

CONDITIONS: Hemostasis

STUDY DESIGN:
Intervention Model Description: 60 patients, randomized into one of three arms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Full Inflation (Other): 100% TR Band inflation relative to recommended inflation with 15-18 cc air injected in TR band bladder
  Interventions: Device: hm-P bandage
- Mid Inflation (Other): 75% TR Band inflation relative to recommended inflation with 11-14 cc air injected in TR band bladder
  Interventions: Device: hm-P bandage
- Low Inflation (Other): 50% TR Band inflation relative to recommended inflation with 8-9 cc air injected in TR band bladder
  Interventions: Device: hm-P bandage

INTERVENTIONS:
Device: hm-P bandage — hm-P bandage will be placed over the puncture site with the TR band positioned over the hemostatic bandage. The TR band will then be inflated per device specific instructions and to the group instructions. The arterial sheath will be removed from the body with slight device rotation.

SUMMARY:
Clinical randomized study to evaluate the effect of using a hydrophobically modified polysaccharide (hm-P) bandage

DETAILED DESCRIPTION:
The study will evaluate the clinical performance (e.g. hemostatic and patient outcomes) of this hm-P bandage by using an earlier time for removal of the bandage (e.g. 60 minutes) than the current standard of care (e.g. 90-180 minutes) while also reducing the inflated pressure of the band, and hence the compressive force put on the wrist of the patient, in increments of the % of inflation as per current protocol, with N=20 @ 100%, N=20 @ 75%, & N=20 @ 50%. This study will be completed while maintaining vascular integrity and patency through visualization in patients undergoing angiographic procedures via anticoagulated, percutaneous radial arterial cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Current patients who are undergoing diagnostic and interventional coronary/vascular angiography via a transradial approach with or without planned coronary or peripheral intervention.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis | 60 minutes
  Significant change in time to hemostasis
Compressive Force | 60 minutes
  Change in the compressive force onto the access site

SECONDARY OUTCOMES:
Radial Artery | immediately after hemostasis
  Evaluation of the radial artery post hemostasis by visual or reverse Barbeau test

CONTACTS AND LOCATIONS:
Overall Officials: Varinder Singh, MD, Principal Investigator — Northwell Health
Locations (1):
- Lenox Hill Hospital - Northwell Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No